CLINICAL TRIAL: NCT05535582
Title: Association of Clinical, Laboratory and Imaging Biomarkers With the Occurrence of Acute Myocardial Infraction in Patients Without Standard Modifiable Risk Factors (The Beyond-SMuRFs Study)
Brief Title: Biomarkers Predicting Acute Myocardial Infraction in Patients Without Standard Modifiable Risk Factors
Acronym: BeyondSMuRFs
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Dimitrios Moysidis, Cardiology Fellow, Aristotle University Of Thessaloniki
Other Study IDs: 64000-20/4/2022
Record Dates: First submitted 2022-09-03; First posted 2022-09-10 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases; Acute Myocardial Infarction; Acute Coronary Syndrome; Metabolic Disturbance
Keywords: Standard modifiable risk factors; Acute Myocardial Infarction; Acute Coronary Syndrome; Clinical Profile; Laboratory Biomarkers; Echocardiographic biomarkers
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — blood chemistry test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with SMuRFs: Patients with acute myocardial infraction with a history of at least one standard modifiable risk factor (SMuRF; smoking, diabetes mellitus, dyslipidemia, hypertension)
  Interventions: Diagnostic Test: Investigation of clinical, laboratory and imaging profile
- SMuRF-less Patients: Patients with acute myocardial infraction without history of any SMuRF
  Interventions: Diagnostic Test: Investigation of clinical, laboratory and imaging profile

INTERVENTIONS:
Diagnostic Test: Investigation of clinical, laboratory and imaging profile — Complete and comprehensive medical interview will be conducted in each eligible patient after revascularization. In addition, patient's laboratory data will be recorded on admission and during hospitalization. Furthermore, each patient will undergo a full echocardiographic examination with a specific protocol.

SUMMARY:
Coronary heart disease (CHD) is the leading cause of mortality worldwide. Every year, millions of people suffer its most adverse manifestation, an acute myocardial infraction (AMI). The majority of these patients present at least one of the standard modifiable risk factors (SMuRFs). These include smoking, hypertension, dyslipidemia, and diabetes mellitus (DM). However, emerging scientific evidence recognizes a clinically significant proportion of patients presenting with life-threatening AMI without any SMuRF (SMuRF-less patients). This proportion of patients with ACS without SMuRF appears to be increasing during the last two decades and has recently been reported as high as 20% (of total AMIs). To date, there are no scientific data capable of highlighting specific risk factors-biomarkers responsible for the development of AMIs SMuRF-less patients. Therefore, two groups of patients with AMI (with SMuRFs vs SMuRF-less) will be compared regarding their clinical, laboratory and imaging (echocardiographic and angiographic) profile, and possible predictive factors leading to SMuRF-less AMI will be evaluated. On the basis of the above, the aim is to prospectively analyze a cohort of well-characterized patients with AMI. The rationale of the study is to investigate potential correlations between metabolic profile of patients and SMuRF-less AMI. This could lead to the development of predictive risk stratification algorithms for patients without SMuRFs and coronary artery disease.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of mortality worldwide. Every year, millions of people suffer its most adverse manifestation, an acute myocardial infraction (AMI). The majority of these patients present at least one of the standard modifiable risk factors (SMuRFs). These include smoking, hypertension, dyslipidemia, and diabetes mellitus (DM). However, emerging scientific evidence recognizes a clinically significant proportion of patients presenting with life-threatening AMI without any SMuRF (SMuRF-less patients). This proportion of patients with ACS without SMuRF appears to be increasing during the last two decades and has recently been reported as high as 20% (of total AMIs). To date, there are no scientific data capable of highlighting specific risk factors-biomarkers responsible for the development of AMIs SMuRF-less patients.

Concurrently, it has been shown that atherogenesis, as well as the subsequent inflammatory processes that can lead to AMI, are not only closely related to dyslipidemia, hypertension, DM and smoking, but also to pro-inflammatory cytokines and proteins (such as Lipoprotein a [LPa], interleukin 6 [IL-6]) and other indicators of inflammation, such as soluble urokinase plasminogen activator receptor (suPAR). This could render these biomarkers potential risk factors for the occurence of AMI. Furthermore, clinical entities, such as various autoimmune and collagen diseases (e.g. rheumatoid arthritis), as well as psychiatric syndromes (such as depression) have been associated with an increased risk of atherosclerotic disease. In addition, newer techniques and measurements in trans-thoracic echocardiography, such as GLS (Global Longitudinal peak systolic strain) and Myocardial Work have been linked to "silent" myocardial ischemia and -there is emerging evidence indicating that they- might predict future cardiovascular events. Therefore, the two groups of patients (with SMuRFs vs SMuRF-less) will be compared regarding their clinical, basic and advanced laboratory, and imaging fingerprints for the assessment of predictive factors leading to SMuRF-less AMIs. On the basis of the above, the aim is to prospectively analyze a cohort of well-characterized patients with AMI. The rationale of the study is to investigate potential correlations between clinical, laboratory and imaging profile of patients and SMuRF-less AMI. This could lead to the development of predictive risk stratification algorithms for patients without SMuRFs and coronary artery disease.

Patients will be enrolled in two academic hospitals and a general military hospital in Thessaloniki, Greece. A complete and comprehensive medical interview will be conducted in each eligible patient after revascularization. From this interview, the following demographic and clinical information will be obtained: age, sex, contact information, exact symptoms and disease history, detailed medical history, diagnostic and therapeutic interventions performed in the past and medication received. In addition, the patient's laboratory data will be recorded on admission and during hospitalization. These will include: complete blood count, biochemical control, coagulation mechanism control, hormonal control, HbA1c, NTproBNP, HsTnT on admission, higher-peak value of HsTnT, and NTproBNP, and LPa, IL-6, suPAR levels on admission. Furthermore, each patient will undergo a full echocardiographic examination with a specific protocol that includes specialized and modern measurements such as Global Longitudinal Strain (GLS) of the left ventricle and the rest heart cavities, as well as non-invasive calculation of myocardial work of the left ventricle (Global Constructive Work, Global Wasted Work, Global Work Index, Global Work Efficiency; Myocardial Work). Univariate and multivariate analysis with linear and logistic regression models will be used to investigate independent prognostic factors contributing to the occurrence of SMuRF-less AMIs. The potential application in daily clinical practice of a derived clinical predictive model-algorithm, possibly including a clinical, laboratory and echocardiographic biomarkers, will contribute to the early prognosis and personalized prevention of such a particular category of AMIs.

ELIGIBILITY:
Inclusion Criteria:

* Age >25 years
* Hospitalization for acute myocardial infarction (AMI) with or without ST elevation (based on Fourth Universal Definition of Myocardial Infarction)
* Coronary angiography before or after hospitalization for AMI, in which at least one stenosis >50% in a major epicardial coronary artery (left anterior descending artery, left circumflex artery, right coronary artery) or a branch thereof with a diameter of at least 2 mm was observed.

Exclusion Criteria:

* Inability or refusal to provide informed consent
* Age >90 years
* History of hospitalization due to AMI prior to the present AMI
* History of coronary revascularization prior to the present AMI AMI

Exclusion Criteria for SMuRF-less patients group only:

* Known history of hypertension and/or antihypertensive treatment prior to AMI
* Use of tobacco products on a systematic basis for up to <60 months (5 years) before AMI
* History of diabetes mellitus type 1 or 2 and/or treatment with antidiabetic tablets or insulin before AMI or diagnosis of diabetes mellitus based on HbA1c during AMI hospitalization
* Known hypercholesterolemia (total chol >200 mg/dl / LDLc >150 mg/dl) or treatment with statins or PCSK9is, before AMI

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >25years old presenting with acute myocardial infraction with or without ST elevation within the previous 4 weeks, with at least one angiographically-testified stenosis>50% in a major epicardial coronary artery
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Clinical, laboratory and imaging biomarkers associated with SMuRF-less myocardial infraction | 2 years
  Identification of differences in the prevalence of clinical features, or/and differences in the levels of laboratory and echocardiographic biomarkers between SMuRF-less myocardial infractions and myocardial infractions in patients with SMuRFs. Each parameter/biomarker will be compared between the two groups and therefore assessments are of the same unit of measurement (e.g. difference in BMI between SMuRF-less patients and patients with SMuRFs or difference in the percentage of history of autoimmune diseass between SMuRF-less patients and patients with SMuRFs or difference in serum levels of Lipoprotein a between these two groups)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Giannopoulos, Associate Professor, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Hippokration General University Hospital of Thessaloniki, Thessaloniki, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moysidis DV, Daios S, Anastasiou V, Liatsos AC, Papazoglou AS, Karagiannidis E, Kamperidis V, Makedou K, Thisiadou A, Karalazou P, Papadakis M, Savopoulos C, Ziakas A, Giannakoulas G, Vassilikos V, Giannopoulos G. Association of clinical, laboratory and imaging biomarkers with the occurrence of acute myocardial infarction in patients without standard modifiable risk factors - rationale and design of the "Beyond-SMuRFs Study". BMC Cardiovasc Disord. 2023 Mar 23;23(1):149. doi: 10.1186/s12872-023-03180-4. PMID 36959584